CLINICAL TRIAL: NCT01762566
Title: Randomized Double-Blind Placebo-Controlled Trial (Wheat vs Placebo) in Wheat Sensitive Patients for Evaluation of Bio-Markers of a Single Referred Symptom (Bloating & Swelling)
Brief Title: Bioelectrical Impedance Analysis of Not-celiac Wheat Sensitivity Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ACPM02
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Not-celiac Gluten (Wheat) Sensitivity
Keywords: Not-celiac gluten (wheat) sensitivity; Bioelectrical impedance analysis; Bloating; Swelling
MeSH Terms: conditions — Hypersensitivity | interventions — Flour; Xylose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wheat (Active Comparator): wheat is administered blindly versus placebo in capsules once
  Interventions: Dietary Supplement: wheat; Dietary Supplement: xylose
- xylose (Placebo Comparator): placebo (xylose) will be administered blindly versus wheat in capsules once
  Interventions: Dietary Supplement: wheat; Dietary Supplement: xylose

INTERVENTIONS:
Dietary Supplement: wheat — wheat is administered blindly versus placebo in capsules once
Dietary Supplement: xylose — placebo (xylose) will be administered blindly versus wheat in a capsule once

SUMMARY:
Aim of the investigators' study is to evaluate one of the symptoms described by patients affected with the so-called "not-celiac wheat sensitivity" (NCWS). NCWS patients may be defined as ones, neither celiac or allergic to wheat, who develop symptoms following wheat consumption and improve on Gluten Free Diet (GFD). Among these, patients often report the appearance of bloating and abdominal pain, and, sometimes, swelling of fingers and face, shortly after ingestion of wheat. They also refer that swelling tends to last for some hours and then to disappear on GFD. To our knowledge, this disorder has never been investigated neither proved.

For the investigators' research, the investigators selected adult patients, both genders, affected with NCWS. Diagnostic criteria include: 1) symptoms disappearance on GFD, 2) testing negative for celiac disease [anti-tTG and EMA, and with biopsy Marsh 0-1] and wheat allergy [serum specific IgE for wheat], 3) positive response to a double-blind placebo-controlled challenge (DBPC) with wheat or placebo.

Patients will be recruited among subjects referring, as outpatients, to the Department of Internal Medicine, 'Giovanni Paolo II' Hospital of Sciacca (Agrigento), and of Internal Medicine of the University of Palermo, from January 2012 to October 2013. The investigators will include patients referring for functional dyspepsia and/or irritable bowel syndrome (IBS)-like symptoms. All recruited patients must report body's swelling immediately after wheat ingestion. In all recruited patients, NCWS diagnosis was posed during the previous years, according to the above mentioned criteria.

Patients, all on GFD for at least 30 days, will undergo to another DBPC with wheat or placebo (xylose), performed by administering capsules coded as A or B containing wheat or xylose, respectively. Capsules A or B will be administered once, and then, after 1 week of washout, patients received the other capsules, given once too. Before and 2 hours after every challenge, patients will undergo a complete medical examination (measurement of body weight, height, body mass index [BMI], waist circumference, diameter of thighs, legs, arms, and fingers), and we will perform bioelectrical impedance analysis and collect blood sampling, for identification of possible markers (bioelectrical, immunologic, hormonal, etc) that may help to demonstrate and explain mechanisms of examined symptom.

DETAILED DESCRIPTION:
Gluten is the most important protein component of some grains, notably wheat, rye, and barley, which are the basis for a variety of wheat-derived alimentary products consumed throughout the world (bread, pasta, pizza etc). However the "engineering" of gluten-containing grains created the conditions for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including celiac disease, wheat allergy and gluten sensitivity, that, combined, seems to affect about 10% of the general population. The frequency of not-celiac gluten sensitivity is however still unknown, even though it is possible that this condition have been undiagnosed and under-diagnosed by the physicians for a long time. The immune responsiveness to wheat antigens represents a complex process, and its establishment and maintenance are not completely elucidated. The most frequent diseases caused by wheat ingestion are T cell-mediated disorders, i.e. celiac disease and immunoglobulin E (IgE)-mediated allergic reactions. However, besides celiac disease and wheat allergy, there are cases of gluten reactions in which neither autoimmune nor IgE-mediated allergic mechanisms are involved. These are generally defined as gluten sensitivity. Some subjects, who experience symptoms when eating gluten-containing products and show improvement when following a gluten-free diet, may have gluten sensitivity instead of celiac disease or wheat allergy. Gluten sensitivity patients are unable to tolerate gluten and develop an adverse reaction when eating gluten, that, usually, and differently from celiac disease, does not lead to small intestinal damage. Gastrointestinal symptoms in gluten sensitivity patients may resemble those associated with celiac disease, but the overall clinical picture is generally less severe and is not accompanied by the occurrence of autoantibodies (i.e. anti-tissue transglutaminase, tTG, or anti-endomysium, EMA) or autoimmune disease (i.e. Hashimoto's thyroiditis). Typically, the diagnosis is made by exclusion, and an elimination diet and an "open challenge" (i.e., the monitored reintroduction of gluten-containing foods) are most often used to evaluate whether health improves or worsen with the elimination or reintroduction of gluten in the diet, respectively.

As it is not known what cereals components determine the symptoms in the so called gluten sensitivity patients, we prefer to define this condition as "wheat sensitivity" instead of "gluten sensitivity".

Wheat sensitivity can cause both gastrointestinal and extra-intestinal symptoms; among the latter, the patients often reported body's swelling (hands', fingers', arms' , face's swelling).

This study has two major aims:

1. Evaluation of the effective dependence from the wheat ingestion of the clinical alterations presented by patients with diagnosed gluten sensitivity, with particular attention to abdominal bloating and body's swelling. The study will be done after a period of gluten-free diet (at least 30 days), using a double-blind placebo-controlled challenge with wheat or placebo (xylose), performed by administering capsules coded as A or B containing wheat or xylose, respectively. Capsules A or B will be administered once, and then, after 1 week of washout, the patients received the other capsules, given once too.
2. Before and 2 hours after every challenge, patients will undergo a complete medical examination, and The investigators will perform bioelectrical impedance analysis and collect blood sampling, for identification of possible markers that may be of help to demonstrate and explain the mechanisms of the examined symptom.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both genders, with age between 18-65 years, with gastrointestinal symptoms/signs that improved on a gluten-free diet and worsen on a wheat containing diet
* Patients testing negative for celiac disease (i.e. anti-tTG and EMA negative, and with biopsy Marsh 0-1) and wheat allergy (serum specific IgE for wheat negative)
* gluten sensitivity diagnosis confirmed with a double-blind placebo-controlled challenge with gluten or placebo

Exclusion Criteria:

* Patients diagnosed with celiac disease (positive anti-tTG and/or EMA, and positive histology - (presence of villi atrophy);
* Patients diagnosed with wheat allergy (positive serum specific IgE for wheat)
* Patients suffering from Diabetes Mellitus
* Patients with Inflammatory Bowel Diseases (Crohn's disease or ulcerative colitis)
* Patients with Helicobacter pylori infection and other gastrointestinal infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Symptom evaluation | Change from baseline and at 2 hours
  Symptom evaluation, before and after the challenge, by complete medical examination, with measurement of body weight, height, body mass index (BMI), waist circumference, diameter of thighs, legs, arms, and fingers

SECONDARY OUTCOMES:
Bio-Markers evaluation | Change from baseline and at 2 hours
  Bio-Markers to that may be of help to demonstrate and explain the mechanisms of the examined symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PHD, Principal Investigator — Internal Medicine, Giovanni Paolo II Hospital of Sciacca (Agrigento) and University of Palermo, Palermo, Italy
Locations (2):
- Italy (2):
  - Internal Medicine, "Giovanni Paolo II" Hospital, Sciacca, Agrigento
  - Internal Medicine, University Hospital of Palermo, Palermo, Palermo